CLINICAL TRIAL: NCT01776424
Title: A Randomized Controlled Trial of Rivaroxaban for the Prevention of Major Cardiovascular Events in Patients With Coronary or Peripheral Artery Disease (COMPASS - Cardiovascular OutcoMes for People Using Anticoagulation StrategieS).
Brief Title: Rivaroxaban for the Prevention of Major Cardiovascular Events in Coronary or Peripheral Artery Disease
Acronym: COMPASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Population Health Research Institute (Other); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15786; 2012-004180-43 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Prevention & Control
Keywords: Cardiovascular events; Rivaroxaban; Xarelto; Anticoagulant; Blood thinner; Aspirin; ASA; Coronary artery disease; CAD; Peripheral artery disease; PAD; Artery disease; Coronary artery bypass graft; Stroke; Heart attack; Angina; Arterial vascular disease; Myocardial infarction; MI; Cardiovascular Death; CV Death; Heart disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Stroke; Myocardial Infarction; Angina Pectoris; Heart Diseases | interventions — Rivaroxaban; Aspirin; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants who consented to COMPASS long-term open-label extension (LTOLE) part received open label rivaroxaban 2.5 mg bid and aspirin 100 mg od in LTOLE part and no blinding procedures were applicable to the LTOLE part.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rivaroxaban 2.5mg + Aspirin 100mg (Experimental): Participants received rivaroxaban 2.5 mg twice daily (bid) and aspirin 100 mg once daily (od). All doses were provided in tablet form for oral administration. Participants who did not have a continuous need to take a proton pump inhibitor (PPI), were additionally randomized 1:1 to receive pantoprazole 40 mg (tablet form for oral administration, od) or matching placebo od. Participants who consented to LTOLE part received open label rivaroxaban 2.5 mg bid and aspirin 100 mg od in LTOLE part.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Aspirin; Drug: Pantoprazole; Drug: Pantoprazole placebo
- Rivaroxaban 5mg + Aspirin Placebo (Experimental): Participants received rivaroxaban 5 mg bid and aspirin placebo od. All doses were provided in tablet form for oral administration. Participants who did not have a continuous need to take a PPI, were additionally randomized 1:1 to receive pantoprazole 40 mg (tablet form for oral administration, od) or matching placebo od. Participants who consented to LTOLE part received open label rivaroxaban 2.5 mg bid and aspirin 100 mg od in LTOLE part.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Aspirin placebo; Drug: Pantoprazole; Drug: Pantoprazole placebo
- Rivaroxaban Placebo + Aspirin 100mg (Active Comparator): Participants received rivaroxaban placebo bid and aspirin 100 mg od. All doses were provided in tablet form for oral administration. Participants who did not have a continuous need to take a PPI, were randomized 1:1 to receive pantoprazole 40 mg (tablet form for oral administration, od) or matching placebo od. Participants who consented to LTOLE part received open label rivaroxaban 2.5 mg bid and aspirin 100 mg od in LTOLE part.
  Interventions: Drug: Aspirin; Drug: Rivaroxaban placebo; Drug: Pantoprazole; Drug: Pantoprazole placebo

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Tablet, 2.5 mg, twice daily, oral
  Arms: Rivaroxaban 2.5mg + Aspirin 100mg
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Tablet, 5 mg, twice daily, oral
  Arms: Rivaroxaban 5mg + Aspirin Placebo
Drug: Aspirin — Tablet, 100 mg, once daily, oral
  Arms: Rivaroxaban 2.5mg + Aspirin 100mg; Rivaroxaban Placebo + Aspirin 100mg
Drug: Aspirin placebo — Aspirin matching placebo, once daily, oral
  Arms: Rivaroxaban 5mg + Aspirin Placebo
Drug: Rivaroxaban placebo — Rivaroxaban matching placebo, twice daily, oral
  Arms: Rivaroxaban Placebo + Aspirin 100mg
Drug: Pantoprazole — Tablet, 40 mg, once daily, oral, for participants who were not on a PPI and who were randomized to pantoprazole
Drug: Pantoprazole placebo — Pantoprazole matching placebo, once daily, oral, for participants who were not on a PPI and who were randomized to pantoprazole placebo

SUMMARY:
The primary objectives of this study are:

* To determine whether rivaroxaban 2.5 mg twice daily (bid) + aspirin 100 mg once daily (od) compared with aspirin 100 mg od reduces the risk of a composite of myocardial infarction, stroke, or cardiovascular death in subjects with coronary artery disease (CAD) or peripheral artery disease (PAD);
* To determine whether rivaroxaban 5 mg bid compared with aspirin 100 mg od reduces the risk of a composite of myocardial infarction, stroke or cardiovascular death in subjects with CAD or PAD.

ELIGIBILITY:
Inclusion Criteria:

- Meet criteria for CAD and/or PAD

Subjects with CAD must also meet at least one of the following criteria:

* Age ≥65, or
* Age <65 and documented atherosclerosis or revascularization involving at least 2 vascular beds, or at least 2 additional risk factors

Exclusion Criteria:

* Stroke within 1 month or any history of hemorrhagic or lacunar stroke
* Severe heart failure with known ejection fraction <30% or New York Heart Association (NYHA) class III or IV symptoms
* Estimated glomerular filtration rate (eGFR)<15 mL/min
* Need for dual antiplatelet therapy, other non-aspirin antiplatelet therapy, or oral anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27395 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (443):
- United States (52):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Anaheim, California
  - Laguna Hills, California
  - Northridge, California
  - Palo Alto, California
  - Santa Rosa, California
  - Sylmar, California
  - Torrance, California
  - Norwalk, Connecticut
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Atlantis, Florida
  - Clearwater, Florida
  - Coral Springs, Florida
  - Jacksonville Beach, Florida
  - Largo, Florida
  - New Port Richey, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - Meridian, Idaho
  - Arlington Heights, Illinois
  - Hazel Crest, Illinois
  - Davenport, Iowa
  - West Des Moines, Iowa
  - Crestview Hills, Kentucky
  - Baltimore, Maryland
  - Haverhill, Massachusetts
  - Alpena, Michigan
  - Jackson, Michigan
  - St Louis, Missouri
  - Kalispell, Montana
  - New Brunswick, New Jersey
  - Cortlandt Manor, New York
  - Kingston, New York
  - Saratoga Springs, New York
  - Durham, North Carolina
  - Pinehurst, North Carolina
  - Elyria, Ohio
  - Sandusky, Ohio
  - Toledo, Ohio
  - Doylestown, Pennsylvania
  - Langhorne, Pennsylvania
  - Yardley, Pennsylvania
  - Sioux Falls, South Dakota
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bellevue, Washington
  - Puyallup, Washington
  - Seattle, Washington
  - Spokane, Washington
- Argentina (30):
  - Adrogué, Buenos Aires
  - Bahía Blanca, Buenos Aires
  - Coronel Suárez, Buenos Aires
  - Junín, Buenos Aires
  - La Plata, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Merlo, Buenos Aires
  - Munro, Buenos Aires
  - Quilmes, Buenos Aires
  - Ramos Mejía, Buenos Aires
  - San Martín, Buenos Aires
  - San Nicolás de los Arroyos, Buenos Aires
  - Vicente López, Buenos Aires
  - Zárate, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Ciudad Autón. de Buenos Aires, Ciudad Auton. de Buenos Aires
  - Villa Allende, Córdoba Province
  - Villa María, Córdoba Province
  - Santa Rosa, La Pampa Province
  - Rafaela, Santa Fe Province
  - Rosario, Santa Fe Province
  - Venado Tuerto, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Ciudad Auton. de Buenos Aires
  - Corrientes
  - Córdoba
  - Salta
  - San Juan
  - San Luis
  - Santa Fe
- Australia (16):
  - Bruce, Australian Capital Territory
  - Gosford, New South Wales
  - New Lambton Heights, New South Wales
  - Taree, New South Wales
  - Birtinya, Queensland
  - Brisbane, Queensland
  - Redcliffe, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Hobart, Tasmania
  - Launceston, Tasmania
  - Geelong, Victoria
  - Melbourne, Victoria
  - Prahran, Victoria
  - Murdoch, Western Australia
  - Nedlands, Western Australia
- Belgium (11):
  - Antwerp
  - Bonheiden
  - Bruges
  - Bruxelles - Brussel
  - Charleroi
  - Genk
  - Hasselt
  - Kortrijk
  - Leuven
  - Liège
  - Roeselare
- Brazil (16):
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Uberaba, Minas Gerais
  - Uberlândia, Minas Gerais
  - Campina Grande do Sul, Paraná
  - Curitiba, Paraná
  - Canoas, Rio Grande do Sul
  - Pelotas, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Blumenau, Santa Catarina
  - Campinas, São Paulo
  - Matão, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
  - Votuporanga, São Paulo
  - São Paulo
- Canada (35):
  - Calgary, Alberta
  - Edmonton, Alberta
  - New Westminster, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Brampton, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - Grimsby, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Chicoutimi, Quebec
  - Laval, Quebec
  - Lévis, Quebec
  - Montreal, Quebec
  - Sherbrooke, Quebec
  - Terrebonne, Quebec
  - Thetford-Mines, Quebec
  - Trois-Rivières, Quebec
  - Ontario
  - Québec
- Chile (8):
  - Concepción, Bío-Bío
  - Osorno, Los Lagos Region
  - Valdivia, Los Lagos Region
  - Temuco, Región de la Araucanía
  - Viña del Mar, Región de Valparaíso
  - Providencia, Santiago Metropolitan
  - San Miguel, Santiago Metropolitan
  - Santiago
- China (13):
  - Guangzhou, Guangdong
  - Wudan, Hubei
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Changchun, Jilin
  - Shenyang, Liaoning
  - Xi’an, Shanxi
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Shanghai
- Colombia (13):
  - Barranquilla, Atlántico
  - Manizales, Caldas Department
  - Cartagena, Departamento de Bolívar
  - Montería, Departamento de Córdoba
  - Pasto, Departamento de Nariño
  - Armenia, Quindío Department
  - Pereira, Risaralda Department
  - Bucaramanga, Santander Department
  - Floridablanca, Santander Department
  - Espinal, Tolima Department
  - Cali, Valle del Cauca Department
  - Barranquilla
  - Bogotá
- Czechia (18):
  - Brno
  - České Budějovice
  - Český Krumlov
  - Hodonín
  - Hradec Králové
  - Jablonec nad Nisou
  - Kolín
  - Liberec
  - Olomouc
  - Ostrava
  - Pardubice
  - Prague
  - Slaný
  - Sušice
  - Třebíč
  - Třinec
  - Uherské Hradiště
  - Zlín
- Denmark (9):
  - Aalborg
  - Aarhus N
  - Copenhagen
  - Hellerup
  - Holbæk
  - Hvidovre
  - Kolding
  - København Ø
  - Viborg
- Ecuador (3):
  - Guayaquil, Guayas
  - Quito, Pichincha
  - Quito
- Finland (5):
  - Kuopio
  - Kuusankoski
  - Tampere
  - Turku
  - Vantaa
- France (8):
  - Amiens
  - Clermont-Ferrand
  - Limoges
  - Montpellier
  - Nice
  - Nîmes
  - Paris
  - Saint-Priest-en-Jarez
- Germany (16):
  - Nuremberg, Bavaria
  - Würzburg, Bavaria
  - Bad Homburg, Hesse
  - Frankfurt am Main, Hesse
  - Kassel, Hesse
  - Bielefeld, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Bottrop
  - Frankfurt
  - Hamburg
  - Warendorf
- Hungary (8):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Mosonmagyaróvár
  - Pécs
  - Sopron
  - Szekszárd
  - Székesfehérvár
- Ireland (4):
  - Ballinasloe, Co. Galway
  - Cork
  - Dublin
  - Galway
- Israel (8):
  - Afula
  - Ashkelon
  - Bnei Brak
  - Haifa
  - Holon
  - Nahariya
  - Safed
  - Tel Aviv
- Italy (19):
  - Foggia, Apulia
  - Lecce, Apulia
  - Caserta, Campania
  - Bologna, Emilia-Romagna
  - Forlì Cesena, Emilia-Romagna
  - Ravenna, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Brescia, Lombardy
  - Cremona, Lombardy
  - Pavia, Lombardy
  - Isernia, Molise
  - Catania, Sicily
  - Palermo, Sicily
  - Ancona, The Marches
  - Arezzo, Tuscany
  - Florence, Tuscany
  - Perugia, Umbria
  - Terni, Umbria
- Japan (36):
  - Nagoya, Aichi-ken
  - Toyoake, Aichi-ken
  - Kisarazu, Chiba
  - Matsudo, Chiba
  - Imabari, Ehime
  - Matsuyama, Ehime
  - Kasuga, Fukuoka
  - Kitakyushu, Fukuoka
  - Miyako-gun, Fukuoka
  - Onga-gun, Fukuoka
  - Maebashi, Gunma
  - Onomichi, Hiroshima
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Tomakomai, Hokkaido
  - Kobe, Hyōgo
  - Takarazuka, Hyōgo
  - Kaga, Ishikawa-ken
  - Miura-gun, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Naha, Okinawa
  - Kishiwada, Osaka
  - Takatsuki, Osaka
  - Tokorozawa, Saitama
  - Komatsushimachō, Tokushima
  - Akishima, Tokyo
  - Bunkyo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Shimonoseki, Yamaguchi
  - Chiba
  - Fukuoka
  - Gifu
  - Kumamoto
  - Kyoto
  - Osaka
- Malaysia (5):
  - Batu Caves, Selangor
  - Kedah
  - Kuala Lumpur
  - Kuala Selangor
  - Sungai Buloh Selangor
- Netherlands (26):
  - 's-Hertogenbosch
  - Amsterdam
  - Apeldoorn
  - Arnhem
  - Breda
  - Delft
  - Deventer
  - Doetinchem
  - Drachten
  - Ede
  - Gorinchem
  - Gouda
  - Groningen
  - Heerlen
  - Helmond
  - Hoogeveen
  - Hoorn
  - Leeuwarden
  - Meppel
  - Nijmegen
  - Roermond
  - Roosendaal
  - Rotterdam
  - Sneek
  - Tiel
  - Zwolle
- Philippines (13):
  - Batangas
  - Cebu City
  - City of Muntinlupa
  - Dagupan
  - Dasmariñas
  - Iloilo City
  - Laoag
  - Manila
  - Metro Manila
  - Palawan
  - Pasig
  - Quezon City
  - Tacloban City
- Poland (6):
  - Gdansk
  - Kielce
  - Krakow
  - Lodz
  - Tarnów
  - Wroclaw
- Romania (7):
  - Timișoara, Timiș County
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Târgu Mureş
  - Timișoara
- Russia (6):
  - Barnaul
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Tomsk
  - Zhukovskiy
- Slovakia (5):
  - Bratislava
  - Košice
  - Nitra
  - Prešov
  - Vráble
- South Africa (9):
  - Pinelands, Eastern Cape
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Freestate
  - Johannesburg, Gauteng
  - Cape Town, Western Cape
  - Observatory, Western Cape
  - Pinelands, Western Cape
  - Worcester, Western Cape
  - Somerset West
- South Korea (8):
  - Wŏnju, Gang''weondo
  - Goyang-si, Gyeonggido
  - Seongnam-si, Gyeonggido
  - Jeju City, Jeju-do
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daejeon
  - Seoul
- Sweden (8):
  - Gothenburg
  - Helsingborg
  - Kristianstad
  - Örebro
  - Östersund
  - Skellefteå
  - Stockholm
  - Vällingby
- Lugano, Canton Ticino, Switzerland
- Ukraine (7):
  - Dnipropetrovsk
  - Kharkiv
  - Kiev
  - Lviv
  - Simferopol
  - Vinnitsa
  - Zaporizhzhya
- United Kingdom (14):
  - Belfast, Antrim
  - Londonderry Co. Londonderry, Derry
  - Basildon, Essex
  - Stevenage, Hertfordshire
  - Blackpool, Lancashire
  - Harrow, London
  - Portadown, North Ireland
  - Middlesbrough, North Yorkshire
  - Northampton, Northamptonshire
  - Hardwick, Stockton-on-Tees
  - Nuneaton, Warwickshire
  - West Bromich, West Midlands
  - Wolverhampton, West Midlands
  - Worcester, Worcestershire

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Background] Eikelboom JW, Bosch J, Connolly SJ, Tyrwitt J, Fox KAA, Muehlhofer E, Neumann C, Tasto C, Bangdiwala SI, Diaz R, Alings M, Dagenais GR, Leong DP, Lonn EM, Avezum A, Piegas LS, Widimsky P, Parkhomenko AN, Bhatt DL, Branch KRH, Probstfield JL, Lopez-Jaramillo P, Ryden L, Pogosova N, Keltai K, Keltai M, Ertl G, Stoerk S, Dans AL, Lanas F, Liang Y, Zhu J, Torp-Pedersen C, Maggioni AP, Commerford PJ, Guzik TJ, Vanassche T, Verhamme P, O'Donnell M, Tonkin AM, Varigos JD, Vinereanu D, Felix C, Kim JH, Ibrahim KS, Lewis BS, Metsarinne KP, Aboyans V, Steg PG, Hori M, Kakkar A, Anand SS, Lamy A, Sharma M, Yusuf S. Long-Term Treatment with the Combination of Rivaroxaban and Aspirin in Patients with Chronic Coronary or Peripheral Artery Disease: Outcomes During the Open Label Extension of the COMPASS trial. Eur Heart J Cardiovasc Pharmacother. 2022 Dec 2;8(8):786-795. doi: 10.1093/ehjcvp/pvac023. PMID 35383832
- [Result] Anand SS, Caron F, Eikelboom JW, Bosch J, Dyal L, Aboyans V, Abola MT, Branch KRH, Keltai K, Bhatt DL, Verhamme P, Fox KAA, Cook-Bruns N, Lanius V, Connolly SJ, Yusuf S. Major Adverse Limb Events and Mortality in Patients With Peripheral Artery Disease: The COMPASS Trial. J Am Coll Cardiol. 2018 May 22;71(20):2306-2315. doi: 10.1016/j.jacc.2018.03.008. Epub 2018 Mar 11. PMID 29540326
- [Result] Anand SS, Bosch J, Eikelboom JW, Connolly SJ, Diaz R, Widimsky P, Aboyans V, Alings M, Kakkar AK, Keltai K, Maggioni AP, Lewis BS, Störk S, Zhu J, Lopez-Jaramillo P, O'Donnell M, Commerford PJ, Vinereanu D, Pogosova N, Ryden L, Fox KAA, Bhatt DL, Misselwitz F, Varigos JD, Vanassche T, Avezum AA, Chen E, Branch K, Leong DP, Bangdiwala SI, Hart RG, Yusuf S. Rivaroxaban with or without aspirin in patients with stable peripheral or carotid artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 Nov 10. pii: S0140-6736(17)32409-1. doi: 10.1016/S0140-6736(17)32409-1. PMID:29132880
- [Result] Connolly SJ, Eikelboom JW, Bosch J, Dagenais G, Dyal L, Lanas F, Metsarinne K, O'Donnell M, Dans AL, Ha JW, Parkhomenko AN, Avezum AA, Lonn E, Lisheng L, Torp-Pedersen C, Widimsky P, Maggioni AP, Felix C, Keltai K, Hori M, Yusoff K, Guzik TJ, Bhatt DL, Branch KRH, Cook Bruns N, Berkowitz SD, Anand SS, Varigos JD, Fox KAA, Yusuf S. Rivaroxaban with or without aspirin in patients with stable coronary artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 Nov 10. pii: S0140-6736(17)32458-3. doi: 10.1016/S0140-6736(17)32458-3. PMID:29132879
- [Result] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Result] Bosch J, Eikelboom JW, Connolly SJ, Bruns NC, Lanius V, Yuan F, Misselwitz F, Chen E, Diaz R, Alings M, Lonn EM, Widimsky P, Hori M, Avezum A, Piegas LS, Bhatt DL, Branch KRH, Probstfield JL, Liang Y, Liu L, Zhu J, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Fox KAA, Kakkar A, Parkhomenko AN, Ertl G, Stork S, Keltai K, Keltai M, Ryden L, Dagenais GR, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Ha JW, Tonkin AM, Varigos JD, Lewis BS, Felix C, Yusoff K, Steg PG, Aboyans V, Metsarinne KP, Anand SS, Hart RG, Lamy A, Moayyedi P, Leong DP, Sharma M, Yusuf S. Rationale, Design and Baseline Characteristics of Participants in the Cardiovascular Outcomes for People Using Anticoagulation Strategies (COMPASS) Trial. Can J Cardiol. 2017 Aug;33(8):1027-1035. doi: 10.1016/j.cjca.2017.06.001. Epub 2017 Jun 8. PMID 28754388
- [Result] Braunwald E. An Important Step for Thrombocardiology. N Engl J Med. 2017 Oct 5;377(14):1387-1388. doi: 10.1056/NEJMe1710241. Epub 2017 Aug 27. No abstract available. PMID 28844176
- [Result] Fauchier L, Bisson A, Angoulvant D. Rivaroxaban in Stable Cardiovascular Disease. N Engl J Med. 2018 Jan 26;378(4):395. doi: 10.1056/NEJMc1714934. No abstract available. PMID 29372976
- [Result] Berger JS. Antithrombotic therapy in peripheral artery disease. Lancet. 2018 Jan 20;391(10117):183-184. doi: 10.1016/S0140-6736(17)32847-7. Epub 2017 Nov 10. No abstract available. PMID 29132877
- [Result] Darmon A, Bhatt DL, Elbez Y, Aboyans V, Anand S, Bosch J, Branch KR, Connolly SJ, Dyal L, Eikelboom JW, Fox KAA, Keltai K, Probstfield J, Yusuf S, Abtan J, Sorbets E, Eagle KA, Ducrocq G, Steg PG. External applicability of the COMPASS trial: an analysis of the reduction of atherothrombosis for continued health (REACH) registry. Eur Heart J. 2018 Mar 1;39(9):750-757a. doi: 10.1093/eurheartj/ehx658. PMID 29186454
- [Result] Verheugt FWA. Return of Oral Anticoagulation in Chronic Stable Coronary Disease. Circulation. 2018 Apr 17;137(16):1655-1657. doi: 10.1161/CIRCULATIONAHA.117.032916. No abstract available. PMID 29661947
- [Result] Fox KAA, Eikelboom JW, Anand SS, Bhatt DL, Bosch J, Connolly SJ, Harrington RA, Steg PG, Yusuf S. Anti-thrombotic options for secondary prevention in patients with chronic atherosclerotic vascular disease: what does COMPASS add? Eur Heart J. 2019 May 7;40(18):1466-1471. doi: 10.1093/eurheartj/ehy347. No abstract available. PMID 29945212
- [Result] Sharma M, Hart RG, Smith EE, Bosch J, Yuan F, Casanova A, Eikelboom JW, Connolly SJ, Wong G, Diaz R, Lopez-Jaramillo P, Ertl G, Stork S, Dagenais GR, Lonn EM, Ryden L, Tonkin AM, Varigos JD, Bhatt DL, Branch KR, Probstfield JL, Kim JH, Ha JW, O'Donnell M, Vinereanu D, Fox KA, Liang Y, Liu L, Zhu J, Pogosova N, Maggioni AP, Avezum A, Piegas LS, Keltai K, Keltai M, Cook Bruns N, Berkowitz S, Yusuf S. Rationale, design, and baseline participant characteristics in the MRI and cognitive substudy of the cardiovascular outcomes for people using anticoagulation strategies trial. Int J Stroke. 2019 Apr;14(3):270-281. doi: 10.1177/1747493018784478. Epub 2018 Jul 30. PMID 30058959
- [Result] Kruger PC, Eikelboom JW, Yusuf S. Rivaroxaban with or without aspirin for prevention of cardiovascular disease. Coron Artery Dis. 2018 Aug;29(5):361-365. doi: 10.1097/MCA.0000000000000605. No abstract available. PMID 29346127
- [Result] Ademi Z, Zomer E, Tonkin A, Liew D. Cost-effectiveness of rivaroxaban and aspirin compared to aspirin alone in patients with stable cardiovascular disease: An Australian perspective. Int J Cardiol. 2018 Nov 1;270:54-59. doi: 10.1016/j.ijcard.2018.06.091. Epub 2018 Jun 25. PMID 30220379
- [Result] Bhagirath VC, Eikelboom JW, Anand SS. Low-dose rivaroxaban plus aspirin for the prevention of cardiovascular events: an evaluation of COMPASS. Future Cardiol. 2018 Nov;14(6):443-453. doi: 10.2217/fca-2018-0059. Epub 2018 Nov 12. PMID 30417662
- [Result] Kruger PC, Anand SS, de Vries TAC, Eikelboom JW. Patients with Peripheral Artery Disease in the COMPASS Trial. Eur J Vasc Endovasc Surg. 2018 Dec;56(6):772-773. doi: 10.1016/j.ejvs.2018.08.010. Epub 2018 Sep 10. No abstract available. PMID 30213508
- [Result] Boden WE, Bhatt DL. Will COMPASS Point to a New Direction in Thrombotic Risk Reduction in Patients With Stable Cardiovascular Disease? Circulation. 2018 Aug 28;138(9):858-860. doi: 10.1161/CIRCULATIONAHA.118.035405. No abstract available. PMID 30354448
- [Result] Lamy A, Eikelboom J, Sheth T, Connolly S, Bosch J, Fox KAA, Zhu J, Lonn E, Dagenais G, Widimsky P, Branch KRH, Bhatt DL, Zheng Z, Straka Z, Dagenais F, Kong Y, Marsden T, Lee SF, Copland I, Yusuf S. Rivaroxaban, Aspirin, or Both to Prevent Early Coronary Bypass Graft Occlusion: The COMPASS-CABG Study. J Am Coll Cardiol. 2019 Jan 22;73(2):121-130. doi: 10.1016/j.jacc.2018.10.048. PMID 30654882
- [Result] Sharma M, Hart RG, Connolly SJ, Bosch J, Shestakovska O, Ng KKH, Catanese L, Keltai K, Aboyans V, Alings M, Ha JW, Varigos J, Tonkin A, O'Donnell M, Bhatt DL, Fox K, Maggioni A, Berkowitz SD, Bruns NC, Yusuf S, Eikelboom JW. Stroke Outcomes in the COMPASS Trial. Circulation. 2019 Feb 26;139(9):1134-1145. doi: 10.1161/CIRCULATIONAHA.118.035864. PMID 30667279
- [Result] Coppens M, Weitz JI, Eikelboom JWA. Synergy of Dual Pathway Inhibition in Chronic Cardiovascular Disease. Circ Res. 2019 Feb;124(3):416-425. doi: 10.1161/CIRCRESAHA.118.313141. PMID 30702997
- [Result] Moayyedi P, Eikelboom JW, Bosch J, Connolly SJ, Dyal L, Shestakovska O, Leong D, Anand SS, Stork S, Branch KRH, Bhatt DL, Verhamme PB, O'Donnell M, Maggioni AP, Lonn EM, Piegas LS, Ertl G, Keltai M, Cook Bruns N, Muehlhofer E, Dagenais GR, Kim JH, Hori M, Steg PG, Hart RG, Diaz R, Alings M, Widimsky P, Avezum A, Probstfield J, Zhu J, Liang Y, Lopez-Jaramillo P, Kakkar A, Parkhomenko AN, Ryden L, Pogosova N, Dans A, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik T, Vinereanu D, Tonkin AM, Lewis BS, Felix C, Yusoff K, Metsarinne K, Fox KAA, Yusuf S; COMPASS Investigators. Pantoprazole to Prevent Gastroduodenal Events in Patients Receiving Rivaroxaban and/or Aspirin in a Randomized, Double-Blind, Placebo-Controlled Trial. Gastroenterology. 2019 Aug;157(2):403-412.e5. doi: 10.1053/j.gastro.2019.04.041. Epub 2019 May 2. PMID 31054846
- [Result] Fox KAA, Eikelboom JW, Shestakovska O, Connolly SJ, Metsarinne KP, Yusuf S. Rivaroxaban Plus Aspirin in Patients With Vascular Disease and Renal Dysfunction: From the COMPASS Trial. J Am Coll Cardiol. 2019 May 14;73(18):2243-2250. doi: 10.1016/j.jacc.2019.02.048. PMID 31072566
- [Result] Cairns JA, Eikelboom JW, Shestakovska O, Yusuf S, DeMets D. Monitoring Emerging Data From the COMPASS Trial of an Antithrombotic Agent. J Am Coll Cardiol. 2019 Jun 4;73(21):2769-2772. doi: 10.1016/j.jacc.2019.03.479. No abstract available. PMID 31146821
- [Result] Moayyedi P, Eikelboom JW, Bosch J, Connolly SJ, Dyal L, Shestakovska O, Leong D, Anand SS, Stork S, Branch KRH, Bhatt DL, Verhamme PB, O'Donnell M, Maggioni AP, Lonn EM, Piegas LS, Ertl G, Keltai M, Bruns NC, Muehlhofer E, Dagenais GR, Kim JH, Hori M, Steg PG, Hart RG, Diaz R, Alings M, Widimsky P, Avezum A, Probstfield J, Zhu J, Liang Y, Lopez-Jaramillo P, Kakkar AK, Parkhomenko AN, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Vinereanu D, Tonkin AM, Lewis BS, Felix C, Yusoff K, Metsarinne KP, Fox KAA, Yusuf S; COMPASS Investigators. Safety of Proton Pump Inhibitors Based on a Large, Multi-Year, Randomized Trial of Patients Receiving Rivaroxaban or Aspirin. Gastroenterology. 2019 Sep;157(3):682-691.e2. doi: 10.1053/j.gastro.2019.05.056. Epub 2019 May 29. PMID 31152740
- [Result] Kruger PC, Guzik TJ, Eikelboom JW. How can the results of the COMPASS trial benefit patients with coronary or peripheral artery disease in Poland? Kardiol Pol. 2019 Aug 23;77(7-8):661-669. doi: 10.33963/KP.14855. Epub 2019 May 30. PMID 31144674
- [Result] Branch KR, Probstfield JL, Eikelboom JW, Bosch J, Maggioni AP, Cheng RK, Bhatt DL, Avezum A, Fox KAA, Connolly SJ, Shestakovska O, Yusuf S. Rivaroxaban With or Without Aspirin in Patients With Heart Failure and Chronic Coronary or Peripheral Artery Disease. Circulation. 2019 Aug 13;140(7):529-537. doi: 10.1161/CIRCULATIONAHA.119.039609. Epub 2019 Jun 5. PMID 31163978
- [Result] Darmon A, Sorbets E, Ducrocq G, Elbez Y, Abtan J, Popovic B, Ohman EM, Rother J, Wilson PF, Montalescot G, Zeymer U, Bhatt DL, Steg PG; REACH Registry Investigators. Association of Multiple Enrichment Criteria With Ischemic and Bleeding Risks Among COMPASS-Eligible Patients. J Am Coll Cardiol. 2019 Jul 2;73(25):3281-3291. doi: 10.1016/j.jacc.2019.04.046. PMID 31248549
- [Result] Anand SS, Eikelboom JW, Dyal L, Bosch J, Neumann C, Widimsky P, Avezum AA, Probstfield J, Cook Bruns N, Fox KAA, Bhatt DL, Connolly SJ, Yusuf S; COMPASS Trial Investigators. Rivaroxaban Plus Aspirin Versus Aspirin in Relation to Vascular Risk in the COMPASS Trial. J Am Coll Cardiol. 2019 Jul 2;73(25):3271-3280. doi: 10.1016/j.jacc.2019.02.079. PMID 31248548
- [Result] Fox KAA, Metra M, Morais J, Atar D. The myth of 'stable' coronary artery disease. Nat Rev Cardiol. 2020 Jan;17(1):9-21. doi: 10.1038/s41569-019-0233-y. Epub 2019 Jul 29. PMID 31358978
- [Result] de Vries TI, Eikelboom JW, Bosch J, Westerink J, Dorresteijn JAN, Alings M, Dyal L, Berkowitz SD, van der Graaf Y, Fox KAA, Visseren FLJ. Estimating individual lifetime benefit and bleeding risk of adding rivaroxaban to aspirin for patients with stable cardiovascular disease: results from the COMPASS trial. Eur Heart J. 2019 Dec 7;40(46):3771-3778a. doi: 10.1093/eurheartj/ehz404. PMID 31504399
- [Result] Eikelboom JW, Connolly SJ, Bosch J, Shestakovska O, Aboyans V, Alings M, Anand SS, Avezum A, Berkowitz SD, Bhatt DL, Cook-Bruns N, Felix C, Fox KAA, Hart RG, Maggioni AP, Moayyedi P, O'Donnell M, Ryden L, Verhamme P, Widimsky P, Zhu J, Yusuf S. Bleeding and New Cancer Diagnosis in Patients With Atherosclerosis. Circulation. 2019 Oct 29;140(18):1451-1459. doi: 10.1161/CIRCULATIONAHA.119.041949. Epub 2019 Sep 12. PMID 31510769
- [Result] Perera KS, Ng KKH, Nayar S, Catanese L, Dyal L, Sharma M, Connolly SJ, Yusuf S, Bosch J, Eikelboom JW, Hart RG. Association Between Low-Dose Rivaroxaban With or Without Aspirin and Ischemic Stroke Subtypes: A Secondary Analysis of the COMPASS Trial. JAMA Neurol. 2020 Jan 1;77(1):43-48. doi: 10.1001/jamaneurol.2019.2984. PMID 31524941
- [Result] Eikelboom JW, Bosch JJ, Connolly SJ, Shestakovska O, Dagenais GR, Hart RG, Leong DP, O'Donnell M, Fox KAA, Bhatt DL, Cairns JA, Tasto C, Berkowitz SD, Cook Bruns N, Muehlhofer E, Diaz R, Maggioni AP, Yusuf S. Major Bleeding in Patients With Coronary or Peripheral Artery Disease Treated With Rivaroxaban Plus Aspirin. J Am Coll Cardiol. 2019 Sep 24;74(12):1519-1528. doi: 10.1016/j.jacc.2019.07.065. PMID 31537259
- [Result] Wurtz M, Olesen KKW, Thim T, Kristensen SD, Eikelboom JW, Maeng M. External applicability of the COMPASS trial: the Western Denmark Heart Registry. Eur Heart J Cardiovasc Pharmacother. 2019 Oct 1;5(4):192-199. doi: 10.1093/ehjcvp/pvz013. PMID 30916315
- [Result] Vanassche T, Verhamme P, Anand SS, Shestakovska O, Fox KA, Bhatt DL, Avezum A, Alings M, Aboyans V, Maggioni AP, Widimsky P, Berkowitz SD, Yusuf S, Connolly SJ, Eikelboom JW, Bosch J. Risk factors and clinical outcomes in chronic coronary and peripheral artery disease: An analysis of the randomized, double-blind COMPASS trial. Eur J Prev Cardiol. 2020 Feb;27(3):296-307. doi: 10.1177/2047487319882154. Epub 2019 Oct 15. PMID 31615291
- [Result] Cowie MR, Lamy A, Levy P, Mealing S, Millier A, Mernagh P, Cristeau O, Bowrin K, Briere JB. Health economic evaluation of rivaroxaban in the treatment of patients with chronic coronary artery disease or peripheral artery disease. Cardiovasc Res. 2020 Sep 1;116(11):1918-1924. doi: 10.1093/cvr/cvz278. PMID 31807773
- [Result] Welsh RC, Peterson ED, De Caterina R, Bode C, Gersh B, Eikelboom JW. Applying contemporary antithrombotic therapy in the secondary prevention of chronic atherosclerotic cardiovascular disease. Am Heart J. 2019 Dec;218:100-109. doi: 10.1016/j.ahj.2019.09.006. Epub 2019 Oct 23. PMID 31715433
- [Result] Schiele F, Puymirat E, Ferrieres J, Simon T, Fox KAA, Eikelboom J, Danchin N; FAST-MI investigators. The FAST-MI 2005-2010-2015 registries in the light of the COMPASS trial: The COMPASS criteria applied to a post-MI population. Int J Cardiol. 2019 Mar 1;278:7-13. doi: 10.1016/j.ijcard.2018.11.138. Epub 2018 Dec 3. PMID 30538057
- [Result] Bainey KR, Welsh RC, Connolly SJ, Marsden T, Bosch J, Fox KAA, Steg PG, Vinereanu D, Connolly DL, Berkowitz SD, Foody JM, Probstfield JL, Branch KR, Lewis BS, Diaz R, Muehlhofer E, Widimsky P, Yusuf S, Eikelboom JW, Bhatt DL; COMPASS Investigators. Rivaroxaban Plus Aspirin Versus Aspirin Alone in Patients With Prior Percutaneous Coronary Intervention (COMPASS-PCI). Circulation. 2020 Apr 7;141(14):1141-1151. doi: 10.1161/CIRCULATIONAHA.119.044598. Epub 2020 Mar 17. PMID 32178526
- [Result] Liang Y, Zhu J, Liu L, Anand SS, Connolly SJ, Bosch J, Guzik TJ, O'Donnell M, Dagenais GR, Fox KA, Shestakovska O, Berkowitz SD, Muehlhofer E, Keller L, Yusuf S, Eikelboom JW; COMPASS Investigators. Efficacy and safety of rivaroxaban plus aspirin in women and men with chronic coronary or peripheral artery disease. Cardiovasc Res. 2021 Feb 22;117(3):942-949. doi: 10.1093/cvr/cvaa100. PMID 32289159
- [Result] Bhatt DL, Eikelboom JW, Connolly SJ, Steg PG, Anand SS, Verma S, Branch KRH, Probstfield J, Bosch J, Shestakovska O, Szarek M, Maggioni AP, Widimsky P, Avezum A, Diaz R, Lewis BS, Berkowitz SD, Fox KAA, Ryden L, Yusuf S; COMPASS Steering Committee and Investigators. Role of Combination Antiplatelet and Anticoagulation Therapy in Diabetes Mellitus and Cardiovascular Disease: Insights From the COMPASS Trial. Circulation. 2020 Jun 9;141(23):1841-1854. doi: 10.1161/CIRCULATIONAHA.120.046448. Epub 2020 Mar 28. PMID 32223318
- [Result] Steffel J, Eikelboom JW, Anand SS, Shestakovska O, Yusuf S, Fox KAA. The COMPASS Trial: Net Clinical Benefit of Low-Dose Rivaroxaban Plus Aspirin as Compared With Aspirin in Patients With Chronic Vascular Disease. Circulation. 2020 Jul 7;142(1):40-48. doi: 10.1161/CIRCULATIONAHA.120.046048. Epub 2020 May 21. PMID 32436455
- [Result] Sharma M, Hart RG, Smith EE, Bosch J, Eikelboom JW, Connolly SJ, Dyal L, Reeh KW, Casanova A, Diaz R, Lopez-Jaramillo P, Ertl G, Stork S, Dagenais GR, Lonn EM, Ryden L, Tonkin AM, Varigos JD, Bhatt DL, Branch KRH, Probstfield JL, Kim JH, O'Donnell M, Vinereanu D, A A Fox K, Liang Y, Liu L, Zhu J, Pogosova N, Maggioni AP, Avezum A, Piegas LS, Keltai K, Keltai M, Berkowitz SD, Yusuf S. Rivaroxaban for Prevention of Covert Brain Infarcts and Cognitive Decline: The COMPASS MRI Substudy. Stroke. 2020 Oct;51(10):2901-2909. doi: 10.1161/STROKEAHA.120.029762. Epub 2020 Sep 21. PMID 32951537
- [Result] Kaplovitch E, Eikelboom JW, Dyal L, Aboyans V, Abola MT, Verhamme P, Avezum A, Fox KAA, Berkowitz SD, Bangdiwala SI, Yusuf S, Anand SS. Rivaroxaban and Aspirin in Patients With Symptomatic Lower Extremity Peripheral Artery Disease: A Subanalysis of the COMPASS Randomized Clinical Trial. JAMA Cardiol. 2021 Jan 1;6(1):21-29. doi: 10.1001/jamacardio.2020.4390. PMID 32997098
- [Result] Guzik TJ, Ramasundarahettige C, Pogosova N, Lopez-Jaramillo P, Dyal L, Berkowitz SD, Muehlhofer E, Bhatt DL, Fox KAA, Yusuf S, Eikelboom JW. Rivaroxaban Plus Aspirin in Obese and Overweight Patients With Vascular Disease in the COMPASS Trial. J Am Coll Cardiol. 2021 Feb 9;77(5):511-525. doi: 10.1016/j.jacc.2020.11.061. PMID 33538248
- [Result] Sen J, Tonkin A, Varigos J, Fonguh S, Berkowitz SD, Yusuf S, Verhamme P, Vanassche T, Anand SS, Fox KAA, Eikelboom JW, Amerena J; COMPASS Trial Investigators. Risk stratification of cardiovascular complications using CHA2DS2-VASc and CHADS2 scores in chronic atherosclerotic cardiovascular disease. Int J Cardiol. 2021 Aug 15;337:9-15. doi: 10.1016/j.ijcard.2021.04.067. Epub 2021 May 3. PMID 33957178
- [Result] Dagenais GR, Dyal L, Bosch JJ, Leong DP, Aboyans V, Berkowitz SD, Bhatt DL, Connolly SJ, Fox KAA, Muehlhofer E, Probstfield JL, Widimsky P, Winkelmann BR, Yusuf S, Eikelboom JW. Cardiovascular consequences of discontinuing low-dose rivaroxaban in people with chronic coronary or peripheral artery disease. Heart. 2021 Jul;107(14):1130-1137. doi: 10.1136/heartjnl-2020-318758. Epub 2021 May 21. PMID 34021038
- [Result] Lamy A, Browne A, Sheth T, Zheng Z, Dagenais F, Noiseux N, Chen X, Bakaeen FG, Brtko M, Stevens LM, Alboom M, Lee SF, Copland I, Salim Y, Eikelboom J; COMPASS Investigators. Skeletonized vs Pedicled Internal Mammary Artery Graft Harvesting in Coronary Artery Bypass Surgery: A Post Hoc Analysis From the COMPASS Trial. JAMA Cardiol. 2021 Sep 1;6(9):1042-1049. doi: 10.1001/jamacardio.2021.1686. PMID 34132753
- [Result] Vanassche T, Verhamme P, Anand SS, Shestakovska O, Leong DP, Fox KAA, Bhatt DL, Avezum A, Alings M, Aboyans V, Maggioni AP, Widimsky P, Muehlhofer E, Berkowitz SD, Yusuf S, Connolly SJ, Eikelboom JW, Bosch J. Low-dose rivaroxaban plus aspirin in patients with polypharmacy and multimorbidity: an analysis from the COMPASS trial. Eur Heart J Cardiovasc Pharmacother. 2022 Aug 11;8(5):462-473. doi: 10.1093/ehjcvp/pvab050. PMID 34191011
- [Result] Eikelboom JW, Bhatt DL, Fox KAA, Bosch J, Connolly SJ, Anand SS, Avezum A, Berkowitz SD, Branch KRH, Dagenais GR, Felix C, Guzik TJ, Hart RG, Maggioni AP, Muehlhofer E, Sharma M, Shestakovska O, Yusuf S. Mortality Benefit of Rivaroxaban Plus Aspirin in Patients With Chronic Coronary or Peripheral Artery Disease. J Am Coll Cardiol. 2021 Jul 6;78(1):14-23. doi: 10.1016/j.jacc.2021.04.083. PMID 34210409
- [Result] Anand SS, Hiatt W, Dyal L, Bauersachs R, Berkowitz SD, Branch KRH, Debus S, Fox KAA, Liang Y, Muehlhofer E, Nehler M, Haskell LP, Patel M, Szarek M, Yusuf S, Eikelboom J, Bonaca MP. Low-dose rivaroxaban and aspirin among patients with peripheral artery disease: a meta-analysis of the COMPASS and VOYAGER trials. Eur J Prev Cardiol. 2022 May 5;29(5):e181-e189. doi: 10.1093/eurjpc/zwab128. PMID 34463737
- [Result] Kaplovitch E, Anand SS. The evolving treatment of peripheral arterial disease: preventing ischaemic events in the post-COMPASS era. Cardiovasc Res. 2019 Oct 1;115(12):e121-e124. doi: 10.1093/cvr/cvz170. No abstract available. PMID 31321405
- [Derived] Lee SF, Ramasundarahettige C, Gerstein HC, McIntyre WF, Eikelboom J, O'Donnell MJ, Zhou Y, Bangdiwala SI, Thabane L. Comparison of total event analysis and first event analysis in relation to heterogeneity in cardiovascular trials. BMC Med Res Methodol. 2025 Jun 9;25(1):159. doi: 10.1186/s12874-025-02593-3. PMID 40490702
- [Derived] Xie F, Yan J, Eikelboom J, Anand S, Muehlhofer E, Pullenayegum E, Wang Y, Avezum A, Bhatt DL, Yusuf S, Bosch J. Health-related quality of life with rivaroxaban plus aspirin vs. aspirin alone in chronic stable cardiovascular disease: Cardiovascular Outcomes for People Using Anticoagulation Strategies (COMPASS) trial. Eur Heart J Open. 2024 Sep 27;4(5):oeae083. doi: 10.1093/ehjopen/oeae083. eCollection 2024 Sep. PMID 39439530
- [Derived] Eikelboom JW, Yi Q, McIntyre WF, Bosch J, Whitlock R, Connolly SJ, Scheier TC, Muehlhofer E, Pap AF, Pocock SJ, Bangdiwala SI. Results of the COMPASS Trial Analyzed Using Win Ratio Compared With Conventional Analytic Approaches. Can J Cardiol. 2024 Nov;40(11):2171-2179. doi: 10.1016/j.cjca.2024.07.002. Epub 2024 Jul 14. PMID 39002945
- [Derived] Leong DP, Bosch J, Bhatt DL, Avezum A, Yuan F, Yusuf S, Eikelboom JW. Impact of Frailty on the Benefits of Dual Pathway Inhibition for the Secondary Prevention of Cardiovascular Events in the COMPASS Randomised Trial. Can J Cardiol. 2025 Jan;41(1):102-111. doi: 10.1016/j.cjca.2024.06.017. Epub 2024 Jun 22. PMID 38914270
- [Derived] Pyne L, Smyth A, Molnar AO, Moayyedi P, Muehlhofer E, Yusuf S, Eikelboom J, Bosch J, Walsh M. The Effects of Pantoprazole on Kidney Outcomes: Post Hoc Observational Analysis from the COMPASS Trial. J Am Soc Nephrol. 2024 Jul 1;35(7):901-909. doi: 10.1681/ASN.0000000000000356. Epub 2024 Apr 11. PMID 38602780
- [Derived] Lamy A, Eikelboom J, Tong W, Yuan F, Bangdiwala SI, Bosch J, Connolly S, Lonn E, Dagenais GR, Branch KRH, Wang WJ, Bhatt DL, Probstfield J, Ertl G, Stork S, Steg PG, Aboyans V, Durand-Zaleski I, Ryden L, Yusuf S; COMPASS Investigators. The Cost-Effectiveness of Rivaroxaban Plus Aspirin Compared with Aspirin Alone in the COMPASS Trial: A US Perspective. Am J Cardiovasc Drugs. 2024 Jan;24(1):117-127. doi: 10.1007/s40256-023-00620-6. Epub 2023 Dec 28. PMID 38153624
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- [Derived] Branch KRH, Probstfield JL, Bosch J, Bhatt DL, Maggioni AP, Muehlhofer E, Avezum A, Widimsky P, Connolly SJ, Yi Q, Shestakovska O, Yusuf S, Eikelboom JW. Total events and net clinical benefit of rivaroxaban and aspirin in patients with chronic coronary or peripheral artery disease: The COMPASS trial. Am Heart J. 2023 Apr;258:60-68. doi: 10.1016/j.ahj.2023.01.008. Epub 2023 Jan 14. PMID 36646196
- [Derived] Smolderen KG, Mena-Hurtado C, Eikelboom JW, Bosch J, Xie F, Ramasundarahettige C, Bhatt DL, Anand SS. Health status and cognitive function for risk stratification in chronic coronary and peripheral artery disease. Eur J Prev Cardiol. 2023 May 9;30(7):535-545. doi: 10.1093/eurjpc/zwac282. PMID 36444513
- [Derived] Gaba P, Bhatt DL, Dagenais GR, Bosch J, Maggioni AP, Widimsky P, Leong D, Fox KAA, Yusuf S, Eikelboom JW; COMPASS Steering Committee and Investigators. Comparison of Investigator-Reported vs Centrally Adjudicated Major Adverse Cardiac Events: A Secondary Analysis of the COMPASS Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2243201. doi: 10.1001/jamanetworkopen.2022.43201. PMID 36409491
- [Derived] Lamy A, Eikelboom J, Tong W, Yuan F, Bangdiwala SI, Bosch J, Connolly S, Lonn E, Dagenais GR, Branch KRH, Wang WJ, Bhatt DL, Probstfield J, Ertl G, Stork S, Steg PG, Aboyans V, Durand-Zaleski I, Ryden L, Yusuf S. The cost-effectiveness of rivaroxaban with or without aspirin in the COMPASS trial. Eur Heart J Qual Care Clin Outcomes. 2023 Aug 7;9(5):502-510. doi: 10.1093/ehjqcco/qcac054. PMID 36001989
- [Derived] Alboom M, Browne A, Sheth T, Zheng Z, Dagenais F, Noiseux N, Brtko M, Stevens LM, Lee SF, Copland I, Power P, Eikelboom J, Lamy A. Conduit selection and early graft failure in coronary artery bypass surgery: A post hoc analysis of the Cardiovascular Outcomes for People Using Anticoagulation Strategies (COMPASS) coronary artery bypass grafting study. J Thorac Cardiovasc Surg. 2023 Mar;165(3):1080-1089.e1. doi: 10.1016/j.jtcvs.2022.05.028. Epub 2022 Jun 2. PMID 35760616
- [Derived] Catanese L, Eikelboom JW, Bosch J, Shestakovska O, Ng K, Nayar S, Perera KS, Shoamanesh A, Sharma M, Hart RG. Oral factor Xa inhibitors and risk of subdural hematoma: COMPASS trial results and meta-analysis. Neurology. 2020 Aug 4;95(5):e480-e487. doi: 10.1212/WNL.0000000000009826. Epub 2020 Jul 10. PMID 32651298
- [Derived] Anand SS, Bosch J, Eikelboom JW, Connolly SJ, Diaz R, Widimsky P, Aboyans V, Alings M, Kakkar AK, Keltai K, Maggioni AP, Lewis BS, Stork S, Zhu J, Lopez-Jaramillo P, O'Donnell M, Commerford PJ, Vinereanu D, Pogosova N, Ryden L, Fox KAA, Bhatt DL, Misselwitz F, Varigos JD, Vanassche T, Avezum AA, Chen E, Branch K, Leong DP, Bangdiwala SI, Hart RG, Yusuf S; COMPASS Investigators. Rivaroxaban with or without aspirin in patients with stable peripheral or carotid artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):219-229. doi: 10.1016/S0140-6736(17)32409-1. Epub 2017 Nov 10. PMID 29132880
- [Derived] Connolly SJ, Eikelboom JW, Bosch J, Dagenais G, Dyal L, Lanas F, Metsarinne K, O'Donnell M, Dans AL, Ha JW, Parkhomenko AN, Avezum AA, Lonn E, Lisheng L, Torp-Pedersen C, Widimsky P, Maggioni AP, Felix C, Keltai K, Hori M, Yusoff K, Guzik TJ, Bhatt DL, Branch KRH, Cook Bruns N, Berkowitz SD, Anand SS, Varigos JD, Fox KAA, Yusuf S; COMPASS investigators. Rivaroxaban with or without aspirin in patients with stable coronary artery disease: an international, randomised, double-blind, placebo-controlled trial. Lancet. 2018 Jan 20;391(10117):205-218. doi: 10.1016/S0140-6736(17)32458-3. Epub 2017 Nov 10. PMID 29132879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 608 centers with randomized participants in 33 countries between 28 Feb 2013 (first patient first visit) and 15 Jun 2021 (last patient last visit of long-term open-label extension part).
Pre-assignment Details: Overall, 29872 participants were screened, of which 2477 participants were screen failures. A total of 27395 participants were randomized to antithrombotic treatment. 17598 participants were randomized to pantoprazole/placebo treatment. 12964 participants joined long-term open-label extension (LTOLE) part.
Period: Antithrombotic Part (Double Blind)
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Started (Randomized to antithrombotic treatment; intention-to-treat analysis set (ITT)) | 9152 | 9117 | 9126
Treated With Antithrombotic Treatment (Safety analysis set (SAF); Antithrombotic treatment: rivaroxaban/placebo and/or study aspirin/placebo) | 9134 | 9109 | 9107
Randomized to Study Pantoprazole/Placebo | 5878 | 5859 | 5861
Completed | 9132 | 9098 | 9102
Not Completed | 20 | 19 | 24
Not completed — Lost to Follow-up | 10 | 8 | 9
Not completed — Withdrawal by Subject | 10 | 11 | 15
Period: LTOLE Part (Open Label)
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Started (LTOLE ITT; All participants were assigned to Rivaroxaban 2.5mg + Aspirin 100mg in LTOLE part; the original arms from Antithrombotic part do not fit any more) | 4399 | 4292 | 4273
Treated in LTOLE Part (LTOLE SAF) | 4379 | 4274 | 4250
Completed (LTOLE part follow-up completed, including death during LTOLE part) | 4320 | 4230 | 4195
Not Completed | 79 | 62 | 78
Not completed — Lost to Follow-up | 6 | 2 | 5
Not completed — Refused | 5 | 2 | 11
Not completed — Missing final visit | 68 | 58 | 62

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set (ITT): included all participants randomized to antithrombotic treatment for the initial study part. The ITT set comprised both participants randomized to pantoprazole/placebo and participants not randomized to pantoprazole/placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg | Total
Number analyzed (Participants) | 9152 | 9117 | 9126 | 27395
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (7.9) | 68.2 (7.9) | 68.2 (8.0) | 68.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2059 | 1972 | 1989 | 6020
  Male | 7093 | 7145 | 7137 | 21375
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 388 | 381 | 376 | 1145
  Hispanic | 1769 | 1751 | 1758 | 5278
  White/Caucasian | 5673 | 5672 | 5682 | 17027
  South Asian | 107 | 102 | 106 | 315
  Other Asian | 956 | 938 | 915 | 2809
  Black/African American | 76 | 94 | 92 | 262
  Other | 183 | 179 | 197 | 559

OUTCOME MEASURES:

1. Primary Outcome: The First Occurrence of the Composite Primary Efficacy Outcome, Myocardial Infarction (MI), Stroke, or Cardiovascular (CV) Death
Description: Count of participants and time from randomization to the first occurrence of the composite primary efficacy outcome, MI, stroke, or CV death were evaluated. Hazard ratios were calculated and reported as statistical analysis.
Time Frame: For each participant, the first occurrence of the composite primary efficacy outcome after randomization up until the global rivaroxaban/aspirin outcomes cut-off date (06 FEB 2017) was considered. The mean time in follow-up until that date was 702 days.
Population: ITT: included all participants randomized to antithrombotic treatment for the initial study part. The ITT set comprised both participants randomized to pantoprazole/placebo and participants not randomized to pantoprazole/placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Rivaroxaban 2.5mg + Aspirin 100mg: Participants received rivaroxaban 2.5 mg twice daily (bid) and aspirin 100 mg once daily (od). All doses were provided in tablet form for oral administration. Participants who did not have a continuous need to take a proton pump inhibitor (PPI), were additionally randomized 1:1 to receive pantoprazole 40 mg (tablet form for oral administration, od) or matching placebo od.
- Rivaroxaban 5mg + Aspirin Placebo: Participants received rivaroxaban 5 mg bid and aspirin placebo od. All doses were provided in tablet form for oral administration. Participants who did not have a continuous need to take a PPI, were additionally randomized 1:1 to receive pantoprazole 40 mg (tablet form for oral administration, od) or matching placebo od.
- Rivaroxaban Placebo + Aspirin 100mg: Participants received rivaroxaban placebo bid and aspirin 100 mg od. All doses were provided in tablet form for oral administration. Participants who did not have a continuous need to take a PPI, were randomized 1:1 to receive pantoprazole 40 mg (tablet form for oral administration, od) or matching placebo od.
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Number analyzed (Participants) | 9152 | 9117 | 9126
Participants | 379 | 448 | 496
Statistical Analysis 1: Comparison: Rivaroxaban 2.5mg + Aspirin 100mg vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.00004, Log Rank — Independent DSMB recommended to stop rivaroxaban/aspirin arms on 06FEB2017. At first interim analysis(~50% events) the log-rank test statistic for one primary comparison had crossed the modified Haybittle-Peto boundary(z=4) consistently over 3 months; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.66 to 0.86] — Stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Rivaroxaban 5mg + Aspirin Placebo vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.11490, Log Rank; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.79 to 1.03] — Stratified Cox proportional hazards model

2. Primary Outcome: The First Occurrence of the Primary Safety Outcome Major Bleeding Based on a Modification of the International Society on Thrombosis and Haemostasis (ISTH) Criteria
Description: Modified ISTH major bleeding is defined as: i) Fatal bleeding, or ii) Symptomatic bleeding in a critical area or organ, such as intraarticular, intracranial, intramuscular with compartment syndrome, intraocular, intraspinal, liver, pancreas, pericardial, respiratory, retroperitoneal, adrenal gland or kidney; or bleeding into the surgical site requiring reoperation, or iii) Bleeding leading to hospitalization (major bleeding also includes presentation to an acute care facility with discharge on the same day).
  Count of participants and time from randomization to the first occurrence of the primary safety outcome major bleeding were evaluated. Hazard ratios were calculated and reported as statistical analysis.
Time Frame: For each participant, the first occurrence of modified ISTH major bleeding after randomization up until the global rivaroxaban/aspirin outcomes cut-off date (06 FEB 2017) was considered. The mean time in follow-up until that date was 702 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Number analyzed (Participants) | 9152 | 9117 | 9126
Participants | 288 | 255 | 170
Statistical Analysis 1: Comparison: Rivaroxaban 2.5mg + Aspirin 100mg vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p < 0.00001, Log Rank; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 1.70, 95% CI 2-sided [1.40 to 2.05] — Stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Rivaroxaban 5mg + Aspirin Placebo vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.00003, Log Rank; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 1.51, 95% CI 2-sided [1.25 to 1.84] — Stratified Cox proportional hazards model

3. Secondary Outcome: The First Occurrence of Myocardial Infarction (MI), Ischemic Stroke, Acute Limb Ischemia (ALI), or Coronary Heart Disease (CHD) Death
Description: Count of participants and time from randomization to the first occurrence of MI, ischemic stroke, ALI, or CHD death were evaluated. Hazard ratios were calculated and reported as statistical analysis.
Time Frame: For each participant, the first occurrence of MI, ALI, or CHD death after randomization up until the global rivaroxaban/aspirin outcomes cut-off date (06 FEB 2017) was considered. The mean time in follow-up until that date was 702 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Number analyzed (Participants) | 9152 | 9117 | 9126
Participants | 329 | 397 | 450
Statistical Analysis 1: Comparison: Rivaroxaban 2.5mg + Aspirin 100mg vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.00001, Log Rank — Nominal p-value; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.63 to 0.83] — Stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Rivaroxaban 5mg + Aspirin Placebo vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.06437, Log Rank — Nominal p-value; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.77 to 1.01] — Stratified Cox proportional hazards model

4. Secondary Outcome: The First Occurrence of MI, Ischemic Stroke, ALI, or Cardiovascular (CV) Death
Description: Count of participants and time from randomization to the first occurrence of MI, ischemic stroke, ALI, or CV death were evaluated. Hazard ratios were calculated and reported as statistical analysis.
Time Frame: For each participant, the first occurrence of MI, ischemic stroke, ALI, or CV death after randomization up until the global rivaroxaban/aspirin outcomes cut-off date (06 FEB 2017) was considered. The mean time in follow-up until that date was 702 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Number analyzed (Participants) | 9152 | 9117 | 9126
Participants | 389 | 453 | 516
Statistical Analysis 1: Comparison: Rivaroxaban 2.5mg + Aspirin 100mg vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.00001, Log Rank — Nominal p-value; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.65 to 0.85] — Stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Rivaroxaban 5mg + Aspirin Placebo vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.03995, Log Rank — Nominal p-value; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.88, 95% CI [0.77 to 0.99] — Stratified Cox proportional hazards model

5. Secondary Outcome: All-cause Mortality
Description: Count of participants and time from randomization to death by all cause were evaluated. Hazard ratios were calculated and reported as statistical analysis.
Time Frame: For each participants, death by any cause after randomization up until the global rivaroxaban/aspirin outcomes cut-off date (06 FEB 2017) was considered. The mean time in follow-up until that date was 702 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg
Number analyzed (Participants) | 9152 | 9117 | 9126
Participants | 313 | 366 | 378
Statistical Analysis 1: Comparison: Rivaroxaban 2.5mg + Aspirin 100mg vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.01062, Log Rank — Nominal p-value; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.71 to 0.96] — Stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Rivaroxaban 5mg + Aspirin Placebo vs Rivaroxaban Placebo + Aspirin 100mg; Test type: Superiority; p = 0.66418, Log Rank — Nominal p-value; Log-rank test (stratified by pantoprazole randomization); Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.84 to 1.12] — Stratified Cox proportional hazards model

6. Other Pre Specified Outcome: The First Occurrence of the Composite Primary Efficacy Outcome, Myocardial Infarction (MI), Stroke, or Cardiovascular (CV) Death in LTOLE Part
Description: Count of participants from COMPASS LTOLE initiation visit to the first occurrence of the composite primary efficacy outcome, MI, stroke, or CV death were evaluated. LTOLE: long-term open-lable extension
Time Frame: For each participant, the first occurrence of the composite primary efficacy outcome after from COMPASS LTOLE initiation visit up until last LTOLE part contact date was considered. The mean time in follow-up was 428 days.
Population: LTOLE ITT: included all participants who completed COMPASS LTOLE initiation visit (LTOLE initiation visit date entered).
Measure: Count of Participants; unit: Participants
Groups:
- LTOLE Part: Rivaroxaban 2.5mg + Aspirin 100mg: Participants who consented to LTOLE part received open label rivaroxaban 2.5 mg bid and aspirin 100 mg od in LTOLE part.
Arm/Group | LTOLE Part: Rivaroxaban 2.5mg + Aspirin 100mg
Number analyzed (Participants) | 12964
Participants | 353

7. Other Pre Specified Outcome: The First Occurrence of the Primary Safety Outcome Major Bleeding Based on a Modification of the International Society on Thrombosis and Haemostasis (ISTH) Criteria in LTOLE Part
Description: Modified ISTH major bleeding is defined as: i) Fatal bleeding, or ii) Symptomatic bleeding in a critical area or organ, such as intraarticular, intracranial, intramuscular with compartment syndrome, intraocular, intraspinal, liver, pancreas, pericardial, respiratory, retroperitoneal, adrenal gland or kidney; or bleeding into the surgical site requiring reoperation, or iii) Bleeding leading to hospitalization (major bleeding also includes presentation to an acute care facility with discharge on the same day).
  Count of participants from COMPASS LTOLE initiation visit to the first occurrence of the primary safety outcome major bleeding was evaluated. LTOLE: long-term open-lable extension
Time Frame: For each participant, the first occurrence of modified ISTH major bleeding from COMPASS LTOLE initiation visit up until 2 days after the last treatment in LTOLE part was considered. The mean time in follow-up was 421 days.
Population: LTOLE SAF: included all participants who completed COMPASS LTOLE initiation visit and who received at least one dose of medication in LTOLE part.
Measure: Count of Participants; unit: Participants
Arm/Group | LTOLE Part: Rivaroxaban 2.5mg + Aspirin 100mg
Number analyzed (Participants) | 12903
Participants | 138

8. Other Pre Specified Outcome: All-cause Mortality in LTOLE Part
Description: Count of participants from COMPASS LTOLE initiation visit to death by all cause were evaluated. LTOLE: long-term open-lable extension
Time Frame: For each participants, death by any cause after COMPASS LTOLE initiation visit up until the the last LTOLE part contact date was considered. The mean time in follow-up until that date was 428 days.
Population: LTOLE ITT: included all participants who completed COMPASS LTOLE initiation visit (LTOLE initiation visit date entered).
Measure: Count of Participants; unit: Participants
Arm/Group | LTOLE Part: Rivaroxaban 2.5mg + Aspirin 100mg
Number analyzed (Participants) | 12964
Participants | 282

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported: from randomization until 2 days after the last antithrombotic study treatment or until LTOLE part initiation visit (including a mean of 478 days in between) for randomized groups (2 years on average); OR from LTOLE initiation visit up until 2 days after the last treatment for LTOLE group (421 days on average). All-Cause Mortality encompasses all death cases until the last contact (2 years on average for randomized groups; 428 days on average for LTOLE group).
Description: During LTOLE part, all participants had stopped randomized treatments and received rivaroxaban 2.5mg+aspirin 100mg od. AEs were collected for safety analysis set (all randomized participants who received at least one dose of antithrombotic study drug). All-Cause Mortality encompasses all deaths in Intent-to-treat analysis set (all randomized participants and/or all who completed LTOLE part initiation visit). 2 participants were treated in LTOLE part never treated in the antithrombotic part.
Groups:
- Rivaroxaban 2.5mg + Aspirin 100mg: Participants received Rivaroxaban 2.5 mg twice daily (bid) and Aspirin 100 mg once daily (od). All doses were provided in tablet form for oral administration.
- Rivaroxaban 5mg + Aspirin Placebo: Participants received Rivaroxaban 5 mg bid and Aspirin placebo od. All doses were provided in tablet form for oral administration.
- Rivaroxaban Placebo + Aspirin 100mg: Participants received Rivaroxaban placebo bid and Aspirin 100 mg od. All doses were provided in tablet form for oral administration.
- LTOLE Rivaroxaban Rivaroxaban 2.5mg + Aspirin 100mg: LTOLE Participants received Rivaroxaban 2.5 mg twice daily (bid) and Aspirin 100 mg once daily (od). All doses were provided in tablet form for oral administration.
Arm/Group | Rivaroxaban 2.5mg + Aspirin 100mg | Rivaroxaban 5mg + Aspirin Placebo | Rivaroxaban Placebo + Aspirin 100mg | LTOLE Rivaroxaban Rivaroxaban 2.5mg + Aspirin 100mg
All-Cause Mortality (participants affected / at risk) | 529/9152 | 566/9117 | 566/9126 | 283/12964
Serious Adverse Events (participants affected / at risk) | 692/9134 | 664/9109 | 630/9107 | 292/12903
Other Adverse Events (participants affected / at risk) | 557/9134 | 529/9109 | 501/9107 | 49/12903
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 2.5mg + Aspirin 100mg (N=9134) | Rivaroxaban 5mg + Aspirin Placebo (N=9109) | Rivaroxaban Placebo + Aspirin 100mg (N=9107) | LTOLE Rivaroxaban Rivaroxaban 2.5mg + Aspirin 100mg (N=12903)
Anaemia (Blood and lymphatic system disorders) | 13 (14) | 10 (11) | 2 (2) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 5 (5) | 10 (10) | 3 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fabry's disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 5 (5) | 6 (6) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 17 (20) | 11 (13) | 7 (9) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmoplegia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden visual loss (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tolosa-Hunt syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular thrombosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (4) | 5 (5) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 3 (3) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallstone ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 6 (7) | 2 (2) | 5 (5) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (7) | 2 (2) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 9 (10) | 8 (9) | 8 (8)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 5 (5) | 10 (10) | 5 (6)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 8 (8) | 14 (14) | 9 (9) | 1 (2)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Omental infarction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Subacute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 9 (9) | 14 (14) | 5 (5) | 2 (2)
Death (General disorders) | 3 (3) | 3 (3) | 7 (7) | 5 (5)
Euthanasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 10 (10) | 5 (6) | 8 (8) | 1 (1)
Accidental death (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Stent-graft endoleak (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site erosion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Lithiasis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 4 (4) | 3 (3) | 2 (2) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 10 (10) | 9 (9) | 12 (12) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 6 (6) | 8 (8) | 9 (9) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 2 (2) | 6 (6) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 7 (7) | 0 (0) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 3 (4) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 9 (9) | 11 (12) | 8 (9) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 5 (5) | 4 (5) | 3 (3) | 2 (2)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear lobe infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 5 (5) | 6 (7) | 4 (4)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 5 (5) | 4 (4) | 2 (2)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 15 (16) | 21 (26) | 22 (22) | 17 (17)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (3) | 4 (4) | 3 (3) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 2 (2) | 3 (4) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 18 (20) | 18 (18) | 17 (17) | 6 (6)
Septic shock (Infections and infestations) | 3 (3) | 7 (7) | 7 (7) | 4 (4)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 17 (19) | 14 (15) | 9 (9) | 7 (7)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral myocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 3 (3) | 8 (9) | 1 (1)
Urosepsis (Infections and infestations) | 9 (9) | 4 (4) | 6 (7) | 8 (9)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 3 (4) | 2 (2) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blindness traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 1 (1) | 2 (2)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 6 (6)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular anastomosis aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Airway burns (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biopsy prostate (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchoscopy (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HIV test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urological examination (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Computerised tomogram thorax (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiogram peripheral (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood electrolytes abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stenotrophomonas test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B core antibody positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiocardiogram (Investigations) | 10 (12) | 9 (9) | 12 (14) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 6 (6) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 5 (5) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (7) | 8 (8) | 0 (0)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 7 (7) | 2 (3)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 6 (6) | 4 (4) | 2 (2)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 8 (9) | 6 (6) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of spermatic cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 7 (7) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (4) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5) | 1 (1) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (18) | 14 (14) | 11 (12) | 8 (8)
Extradural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 10 (10) | 4 (4) | 4 (4)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malignant mesenchymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Central nervous system neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 7 (8) | 5 (5) | 4 (4)
Temporal lobe epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuromuscular pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stereotypy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 6 (6) | 2 (2) | 3 (3) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 8 (8) | 6 (6) | 5 (6) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 2 (2) | 3 (3) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 29 (30) | 22 (22) | 20 (20) | 8 (8)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 7 (7) | 1 (1) | 2 (2) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 8 (9) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11) | 6 (6) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 4 (4) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 4 (4) | 2 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 7 (7) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough variant asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Negative pressure pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (3) | 4 (4) | 5 (5) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Capillaritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy of partner (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia hiatus repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Mole excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ptosis repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glaucoma surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus management (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sigmoidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 2 (3) | 3 (4) | 6 (8) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular graft (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma closure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter management (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renovascular hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atheroembolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban 2.5mg + Aspirin 100mg (N=9134) | Rivaroxaban 5mg + Aspirin Placebo (N=9109) | Rivaroxaban Placebo + Aspirin 100mg (N=9107) | LTOLE Rivaroxaban Rivaroxaban 2.5mg + Aspirin 100mg (N=12903)
Anaemia (Blood and lymphatic system disorders) | 14 (24) | 11 (13) | 9 (11) | 4 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (10) | 12 (16) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 24 (41) | 18 (32) | 18 (27) | 7 (11)
Vertigo (Ear and labyrinth disorders) | 10 (13) | 13 (19) | 15 (19) | 0 (0)
Cataract (Eye disorders) | 12 (12) | 15 (16) | 12 (13) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 10 (13) | 11 (14) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 17 (32) | 10 (20) | 9 (16) | 4 (7)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 12 (23) | 3 (3) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 28 (42) | 18 (30) | 21 (28) | 5 (10)
Constipation (Gastrointestinal disorders) | 26 (33) | 18 (20) | 24 (37) | 0 (0)
Dental caries (Gastrointestinal disorders) | 15 (15) | 12 (13) | 10 (10) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 48 (65) | 58 (79) | 26 (32) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 14 (19) | 12 (20) | 15 (24) | 1 (2)
Gastritis (Gastrointestinal disorders) | 19 (28) | 7 (7) | 13 (21) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 11 (13) | 11 (13) | 6 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (30) | 17 (26) | 14 (21) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 12 (12) | 12 (12) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (9) | 8 (9) | 11 (14) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 16 (17) | 12 (14) | 8 (8) | 1 (1)
Chest discomfort (General disorders) | 5 (5) | 3 (4) | 10 (10) | 0 (0)
Chest pain (General disorders) | 7 (11) | 8 (11) | 10 (10) | 1 (1)
Oedema peripheral (General disorders) | 3 (7) | 7 (8) | 12 (15) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 10 (10) | 8 (9) | 0 (0)
Bronchitis (Infections and infestations) | 14 (15) | 7 (7) | 13 (13) | 0 (0)
Cystitis (Infections and infestations) | 6 (6) | 10 (13) | 7 (7) | 0 (0)
Gastroenteritis (Infections and infestations) | 16 (21) | 10 (10) | 10 (11) | 0 (0)
Herpes zoster (Infections and infestations) | 9 (9) | 15 (15) | 19 (21) | 0 (0)
Influenza (Infections and infestations) | 18 (18) | 14 (16) | 24 (25) | 0 (0)
Nasopharyngitis (Infections and infestations) | 188 (284) | 181 (284) | 195 (289) | 0 (0)
Periodontitis (Infections and infestations) | 12 (13) | 11 (11) | 12 (12) | 0 (0)
Pharyngitis (Infections and infestations) | 8 (8) | 7 (7) | 10 (11) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 37 (42) | 22 (26) | 27 (41) | 2 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 11 (12) | 4 (4) | 3 (3) | 0 (0)
Occult blood positive (Investigations) | 12 (12) | 7 (7) | 3 (4) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 26 (27) | 16 (16) | 28 (28) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (32) | 26 (31) | 30 (36) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (27) | 37 (39) | 25 (27) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 10 (10) | 5 (5) | 6 (6) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (12) | 6 (9) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 14 (18) | 13 (14) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (7) | 10 (10) | 8 (10) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (19) | 8 (10) | 9 (12) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (7) | 8 (8) | 0 (0)
Dizziness (Nervous system disorders) | 25 (41) | 25 (36) | 35 (42) | 2 (3)
Headache (Nervous system disorders) | 20 (31) | 21 (32) | 22 (32) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 8 (9) | 12 (15) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 12 (14) | 4 (4) | 1 (2)
Haematuria (Renal and urinary disorders) | 23 (31) | 15 (25) | 7 (8) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 12 (18) | 11 (13) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 38 (73) | 29 (45) | 24 (29) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (25) | 5 (6) | 5 (5) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 8 (9) | 4 (4) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 17 (23) | 19 (25) | 20 (22) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 49 (86) | 18 (23) | 17 (29) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (27) | 23 (37) | 17 (21) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 12 (22) | 16 (31) | 18 (30) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 11 (13) | 11 (11) | 5 (5) | 1 (2)
Hypertension (Vascular disorders) | 25 (25) | 16 (18) | 11 (11) | 1 (2)

LIMITATIONS AND CAVEATS:
One participant that was included in the Safety Analysis Set in the disclosure after primary completion never took any study drug therefore was corrected in the later analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Global principal investigator (PI) to provide to Bayer for review any proposed Publication/oral presentation relating to Study/Study Drug/Results at least 45 days prior to submission or presentation of the Publication. Abstracts to be provided to Bayer 5 working days before Publication. Bayer may provide comments within the applicable period. Under certain circumstances Bayer may request a further delay of publications to avoid adverse effects on a Bayer patent application.

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT01776424/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT01776424/SAP_003.pdf